CLINICAL TRIAL: NCT00845117
Title: Cultivated Stem Cell Transplantation for the Treatment of Limbal Stem Cell Deficiency
Acronym: LECT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ethisch Comité UZ Antwerpen (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other); European Society of Cataract and Refractive Surgeons (Other); Agentschap voor Innovatie door Wetenschap en Technologie (Other)
Responsible Party: Sponsor-Investigator, Ethisch Comité UZ Antwerpen, Prof. Dr. Marie-Jose Tassignon, University Hospital, Antwerp
Organization: University Hospital, Antwerp (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 7/28/153
Record Dates: First submitted 2009-02-17; First posted 2009-02-18 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2013-06

CONDITIONS: Limbal Stem Cell Deficiency
Keywords: Aniridia,; Steven Johnsons Syndrome,; Ocular burns,; Pterygium
MeSH Terms: conditions — Limbal Stem Cell Deficiency; Aniridia; Stevens-Johnson Syndrome; Pterygium

ARMS (1):
- Limbal Stem Cell Transplant (Experimental): The cornea is debrided of all superficial fibrovascular tissue and the cultivated stem cell graft is glued onto the cornea.
  Interventions: Procedure: Cultivated limbal stem cell graft transplantation

INTERVENTIONS:
Procedure: Cultivated limbal stem cell graft transplantation — A limbal biopsy taken from the contralateral good eye in cases of unilateral disease or from a living related or cadaveric donor in cases of bilateral disease. The limbal stem cells from the biopsy are cultivated until a sheet of cells measuring approximately 12mm in diameter is obtained. This is then ready for transplantation onto the diseased eye.

SUMMARY:
The purpose of this study is to determine whether cultivated stem cell transplantation is effective for the treatment of patients wtih corneal stem cell deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Patients suffering from LSCD IIa and IIb. Those suffering from IIc may be included once inflammation has subsided and cornea can be staged as IIb.
* Absence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial.
* Women of child-bearing potential should use adequate contraception prior to study entry and for the duration of study participation

Exclusion Criteria:

* Subjects who are pregnant or lactating
* Subjects who have sensitivity to drugs that provide local anesthesia
* Subjects suffering from active infection of the external eye
* Medical conditions that prohibit the use of systemic immunosuppression (in cases of allogenic transplantation)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2008-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-06 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | Just before surgery and upto 1 years after surgery
Conjunctivalization | Just before surgery and upto 1 years after surgery
Vascularization | Just before surgery and upto 1 years after surgery
Epithelialization | Just before surgery and upto 1 years after surgery

SECONDARY OUTCOMES:
Prolonged subsequent corneal graft survival time | 1 year post corneal transplant

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Zakaria, MBBS, PhD, Principal Investigator — University Hospital, Antwerp; Carina Koppen, MD, PhD, Principal Investigator — University Hospital, Antwerp; Marie J Tassignon, MD, PhD, Study Director — University Hospital, Antwerp; Zwi Berneman, MD,PhD, Study Chair — University Hospital, Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Edegem, Belgium

REFERENCES:
- [Background] Zakaria N, Koppen C, Van Tendeloo V, Berneman Z, Hopkinson A, Tassignon MJ. Standardized limbal epithelial stem cell graft generation and transplantation. Tissue Eng Part C Methods. 2010 Oct;16(5):921-7. doi: 10.1089/ten.TEC.2009.0634. PMID 19916804